CLINICAL TRIAL: NCT01753167
Title: A Phase II Randomized, Double-blind, Placebo-controlled Trial of MCMV5322A/MCMV3068A for the Prevention of Cytomegalovirus Disease in High-risk Kidney Allograft Recipients
Brief Title: A Study of MCMV5322A/MCMV3068A for the Prevention of Cytomegalovirus Disease in High-Risk Kidney Allograft Recipients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GV28418; 2012-002245-37 (EudraCT Number)
Record Dates: First submitted 2012-12-17; First posted 2012-12-20 (Estimated); Last update posted 2017-03-08 (Actual); Status verified 2017-03

CONDITIONS: Cytomegalovirus Infections
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- MCMV5322A/MCMV3068A (Experimental): Participants will receive a total of four doses of study drug administered by intravenous infusion: at the time of transplantation (Day 1), and at Days 8, 29, and 57. MCMV5322A/MCMV3068A will be tested in this study at 10 milligrams per kilogram (mg/kg) of each component antibody. Thus, at each dose, 10 mg/kg of MCMV5322A and 10 mg/kg of MCMV3068A will be tested (20 mg/kg total).
  Interventions: Drug: MCMV3068A; Drug: MCMV5322A
- Placebo (Placebo Comparator): Participants will receive a total of four doses of placebo matched with MCMV5322A/MCMV3068A administered by intravenous infusion: at the time of transplantation (Day 1), and at Days 8, 29, and 57.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MCMV3068A — Four doses of MCMV3068A (10 mg/kg) administered by intravenous infusion at the time of transplantation (Day 1), and at Days 8, 29, and 57.
  Arms: MCMV5322A/MCMV3068A
Drug: MCMV5322A — Four doses of MCMV5322A (10 mg/kg) administered by intravenous infusion at the time of transplantation (Day 1), and at Days 8, 29, and 57.
  Arms: MCMV5322A/MCMV3068A
Drug: Placebo — Four doses of placebo matched to MCMV5322A/MCMV3068A administered by intravenous infusion at the time of transplantation (Day 1), and at Days 8, 29, and 57.
  Arms: Placebo

SUMMARY:
This is a Phase II, randomized, double-blind, placebo-controlled study designed to assess the safety and clinical activity of multiple intravenous doses of MCMV5322A/MCMV3068A in cytomegalovirus (CMV)-seronegative recipients of a renal transplant from a CMV-seropositive donor, with use of a preemptive approach for prevention of CMV disease. Participants will be randomized into two treatment groups: active or placebo control; both arms will be followed preemptively. The study has a planned enrollment of approximately 120 participants (60 active and 60 placebo).

ELIGIBILITY:
Inclusion Criteria:

* Participant is scheduled to receive a primary or secondary renal allograft from a donor
* Participant is seronegative for CMV and is receiving an allograft from a CMV-seropositive donor
* Female participants of child-bearing age must have a negative pregnancy test result on Day 1, prior to infusion
* For women who are not postmenopausal or surgically sterile (defined as absence of ovaries and/or uterus): agreement to remain completely abstinent or use two methods of contraception at all times

Exclusion Criteria:

* Participant is suspected of having CMV disease
* Participant has received anti-CMV therapy within the 30 days prior to screening (exceptions are the use of acyclovir, valacyclovir, or famciclovir for up to 10 days duration for treatment of acute herpes simplex or herpes zoster or participants receiving acyclovir or valacyclovir at doses to suppress herpes zoster)
* Participants who have received intravenous immunoglobulin (IVIG) within 3 months before transplantation or with expectation of receiving IVIG at time of transplantation or in the 3 months after transplantation
* Participants who have received B cell-depleting therapies (including but not limited to rituximab) within 3 months before transplantation or with the expectation of receiving such therapy at the time of transplantation or in the 3 months after transplantation
* Participant is receiving a multi-organ transplant (e.g., liver or pancreas in addition to kidney)
* Active or chronic hepatic or hepatobiliary disease (including known Gilbert's syndrome) or elevations in a hepatic transaminase or bilirubin >= 2 times upper limits of normal (ULN)
* Participant is unlikely or unwilling to be available for follow-up for the full 24-week duration of the study
* Female participants who are pregnant, plan to become pregnant during the study, or who are breastfeeding
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins or human-derived immunoglobulin preparations; or any constituent of MCMV5322A/MCMV3068A or placebo
* Active treatment for untreated tuberculosis or other infectious conditions that are significant in the judgment of the investigator
* Infection with hepatitis B, hepatitis C or human immunodeficiency virus
* Previous exposure to any investigational agent within 12 weeks or 5 half-lives
* Any other acute or chronic condition, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that, in the opinion of the Principal Investigator, contraindicates the use of an investigational drug or that may affect the interpretation of the results or that renders the participant at high risk for treatment complications
* History of alcoholism or substance abuse within 6 months before screening
* Participant is expected to require treatment or prophylaxis with an antiviral with anti-CMV activity during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2012-12-14 (Actual); Primary Completion 2014-10-15 (Actual); Study Completion 2014-10-15 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Adverse Events | Baseline up to Week 24
Percentage of Participants With CMV Viral Load Greater than or Equal to (>=) 150 Copies per Milliliter (Copies/mL) During the First 12 Weeks After Transplantation | Baseline up to Week 12

SECONDARY OUTCOMES:
Percentage of Participants With CMV Viral Load >= 150 Copies/mL During the First 24 Weeks After Transplantation | Baseline up to Week 24
Time to Detectable CMV Viral Load >=150 Copies/mL | Baseline up to Week 24
Viral Load at the First Detection of CMV DNAemia (>=150 Copies/mL), DNAemia is detection of deoxyribonucleic acid (DNA) | Baseline up to Week 24
Peak Viral Load on or Following First Detection of CMV DNAemia (>=150 Copies/mL) | Baseline up to Week 24
Percentage of Participants who Require Initiation of Pre-emptive Antiviral Therapy During the First 12 Weeks and 24 Weeks After Transplantation | Baseline up to Weeks 12 and 24
Time to Initiation of First use of Preemptive Antiviral Therapy | Baseline up to Week 24
Duration of First use of Preemptive Antiviral Therapy Initiated During the First 12 and 24 Weeks After Transplantation | Baseline up to Weeks 12 and 24
Percentage of Participants With CMV Syndrome or Tissue-Invasive CMV Disease During the First 24 Weeks After Transplantation | Baseline up to Week 24
Percentage of Participants With Change in CMV Serostatus | Baseline up to Week 24
MCMV5322A Serum Concentrations | Up to 24 hours prior to dosing (Day 1) and 1, 4, 24, and 72 hours postdose; predose (0 hours) and 1 hour postdose on Days 8, 29, 57; on Days 43, 58, 64, 71, 78, 85, 113, and 141; at study completion (Day 169)
MCMV3068A Serum Concentrations | Up to 24 hours prior to dosing (Day 1) and 1, 4, 24, and 72 hours postdose; predose (0 hours) and 1 hour postdose on Days 8, 29, 57; on Days 43, 58, 64, 71, 78, 85, 113, and 141; at study completion (Day 169)
Percentage of Participants With Anti-therapeutic Antibodies (ATAs) to MCMV5322A and MCMV3068A | Predose (0 hours) on Days 1, 29, 57; at Days 85, 113, and 141; and at Study Completion (Day 169)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (39):
- United States (15):
  - UCLA; Kidney & Pancreas Transplantation, Los Angeles, California
  - California Inst. of Renal Research, San Diego, California
  - Univ of CA San Francisco; Kidney Transplant Service, San Francisco, California
  - University of Colorado Health Sciences Center; Dept of Medicine, Denver, Colorado
  - Georgetown Uni Hospital; Division of Transplant Surgery, Washington D.C., District of Columbia
  - MedStar Washington Hosp Center, Washington D.C., District of Columbia
  - Emory University, Atlanta, Georgia
  - Georgia Regents University, Augusta, Georgia
  - Henry Ford Health System; Gastroenterology, Detroit, Michigan
  - Washington Uni School of Medicine/Barnes Jewish Hospital; Renal, St Louis, Missouri
  - Erie County Medical Center; Dept. of Nephrology, Buffalo, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Columbia University, New York, New York
  - University of Cincinnati / University of Cincinnati College of Medicine, Cincinnati, Ohio
  - Baylor Univ Medical Center, Dallas, Texas
- Belgium (3):
  - Clin Univ de Bxl Hôpital Erasme, Brussels
  - UZ Gent, Ghent
  - UZ Leuven Gasthuisberg, Leuven
- France (6):
  - Hopital Pellegrin-CHU de Bordeaux; Service de Neurologie, Bordeaux
  - CHU de Nantes; Institut de transplantation urologie-néphrologie, Nantes
  - Hopital Necker, Paris
  - Hopital Rangueil; Gastro Enterologie Et Nutrition, Toulouse
  - Chu De Tours, Tours
  - Hopitaux De Brabois; Nephrologie, Vandœuvre-lès-Nancy
- Germany (4):
  - Universitätsklinikum "Carl Gustav Carus"; Medizinische Klinik III, Dresden
  - Universitätsklinikum Essen Zentrum f.Innere Medizin Abt.Nephrologie, Essen
  - Klinik Johann Wolfgang von Goethe Uni; Zentrum der Inneren Medizin; Medizinische Klinik III, Frankfurt
  - Uniklinikum Heidelberg, Heidelberg
- Oslo Universitetssykehus HF, Rikshospitalet, Oslo, Norway
- Spain (5):
  - Fundació Puigvert, Barcelona, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona
  - Hospital Clinic i Provincial de Barcelona, Barcelona, Barcelona
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - CEIC del Hospital Virgen del Rocío, Seville, Sevilla
- Sweden (3):
  - Sahlgrenska Universitetssjukhuset; Jubileumskliniken, Gothenburg
  - Karolinska University Hospital, Huddinge
  - Akademiska Sjukhuset; Transplantation Surgery, Uppsala
- United Kingdom (2):
  - Royal Free Hospital, London
  - Guys and St Thomas NHS Foundation Trust, Guys Hospital, London

REFERENCES:
- [Derived] Vernooij RW, Michael M, Colombijn JM, Owers DS, Webster AC, Strippoli GF, Hodson EM. Pre-emptive treatment for cytomegalovirus viraemia to prevent cytomegalovirus disease in solid organ transplant recipients. Cochrane Database Syst Rev. 2025 Jan 14;1(1):CD005133. doi: 10.1002/14651858.CD005133.pub4. PMID 39807668
- [Derived] Vernooij RW, Michael M, Ladhani M, Webster AC, Strippoli GF, Craig JC, Hodson EM. Antiviral medications for preventing cytomegalovirus disease in solid organ transplant recipients. Cochrane Database Syst Rev. 2024 May 3;5(5):CD003774. doi: 10.1002/14651858.CD003774.pub5. PMID 38700045
- [Derived] Deng R, Wang Y, Maia M, Burgess T, McBride JM, Liao XC, Tavel JA, Hanley WD. Pharmacokinetics and Exposure-Response Analysis of RG7667, a Combination of Two Anticytomegalovirus Monoclonal Antibodies, in a Phase 2a Randomized Trial To Prevent Cytomegalovirus Infection in High-Risk Kidney Transplant Recipients. Antimicrob Agents Chemother. 2018 Jan 25;62(2):e01108-17. doi: 10.1128/AAC.01108-17. Print 2018 Feb. PMID 29133549
- [Derived] Ishida JH, Patel A, Mehta AK, Gatault P, McBride JM, Burgess T, Derby MA, Snydman DR, Emu B, Feierbach B, Fouts AE, Maia M, Deng R, Rosenberger CM, Gennaro LA, Striano NS, Liao XC, Tavel JA. Phase 2 Randomized, Double-Blind, Placebo-Controlled Trial of RG7667, a Combination Monoclonal Antibody, for Prevention of Cytomegalovirus Infection in High-Risk Kidney Transplant Recipients. Antimicrob Agents Chemother. 2017 Jan 24;61(2):e01794-16. doi: 10.1128/AAC.01794-16. Print 2017 Feb. PMID 27872061